CLINICAL TRIAL: NCT06672770
Title: Investigation of the Effects of Functional Inspiratory Muscle Training on Respiratory Muscle Strength, Functional Exercise Capacity and Cognitive Function in Patients with Multiple Sclerosis
Brief Title: Effect of Functional Inspiratory Muscle Training in Patients with Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mehmet Kaan ALTUNOK, Lecturer, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SelcukU_PT_MS_FIMT-IMT_Resp.01
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Core Muscles; Functional Inspiratory Muscle Training; Multiple Sclerosis; Respiratory Muscles
Keywords: Core muscles; Functional inspiratory muscle training; Multiple sclerosis; Respiratory muscles
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: MS patients will be divided into 3 groups as functional inspiratory muscle training (FIMT) group (n=21), basic inspiratory muscle training (IMT) group (n=21) and Control (CT) group (n=21) by block randomization with the randomization program "https://www.studyrandomizer.com/".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Functional Inspiratory Muscle Training Group (Experimental): The functional inspiratory muscle training (FIMT) group (n=21) will receive basic inspiratory muscle training (IMT) with a device capable of delivering threshold pressure loading (POWERbreathe) for the first four weeks. The first, middle and last sessions of the week will be supervised (face-to-face) and other sessions will be unsupervised (at home, twice a day, totaling 30 minutes). The intensity of inspiratory muscle training will be adjusted to 50-60% of maximal inspiratory pressure and these measurements will be repeated at the beginning of each week and weekly pressure increases will be adjusted. After the first four weeks are completed, then inspiratory muscle training will be combined with exercises at the beginning of the fifth week, and participants will perform supervised in-person FIMT three days per week for four weeks and unsupervised home IMT on the remaining days.
  Interventions: Other: Functional Inspiratory Muscle Training
- Basic Inspiratory Muscle Training Group (Experimental): Basic inspiratory muscle training (IMT) group (n=21) will be given IMT with a device capable of performing threshold pressure loading (POWERbreathe Classic Light Resistance, PowerBreath, IMT Technologies Ltd, Birmingham, UK) for eight weeks. The first day of the week, the middle of the week and the last session will be supervised (face-to-face), and the other sessions will be unsupervised (at home, twice a day, 30 minutes in total). The intensity of inspiratory muscle training will be adjusted to be 50-60% of the maximal inspiratory pressure, and these measurements will be repeated at the beginning of each week and weekly pressure increases will be adjusted.
  Interventions: Other: Basic Inspiratory Muscle Training
- Control Group (No Intervention): Participants in the control group (n=21) will be informed about the benefits of at least 150-300 minutes of moderate intensity or 75-150 minutes of vigorous intensity aerobic physical activity and breathing exercises per week and exercise recommendations will be given. Both daily physical activities and breathing exercises will be monitored with a pre-prepared exercise tracking form. Participants will be called to the laboratory for clinical measurements at the beginning and end of the study.
  Participants in the control group will be taught to do diaphragmatic breathing, thoracic expansion, pursed lip breathing and breath control breathing exercises for 20 minutes a day and will be given as home exercises without supervision, with 1-2 minutes of rest between each exercise.

INTERVENTIONS:
Other: Functional Inspiratory Muscle Training — The functional inspiratory muscle training group will perform basic inspiratory muscle training in the first four weeks of the study and the following exercises with the Powerbreath device in muscle training in the following four weeks:
  1. Diaphragmatic breathing exercises
  2. Warm-up exercises
  3. Trunk strength and lumbopelvic stability exercises
  4. Dynamic trunk exercises
  5. Postural control exercises
  6. Cool-down exercises
  Arms: Functional Inspiratory Muscle Training Group
Other: Basic Inspiratory Muscle Training — The basic inspiratory muscle training group will do muscle training with the POWERbreathe device for eight weeks.
  Arms: Basic Inspiratory Muscle Training Group

SUMMARY:
This study aims to investigate the effects of functional inspiratory muscle training, basic inspiratory muscle training and physical activity in addition to respiratory exercises on respiratory muscle strength, respiratory function, cognition, walking, balance, functional exercise capacity, physical activity, quality of life and core muscles in volunteer Multiple Sclerosis (MS) patients. This study is planned as a prospective, randomized and experimental study.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is an autoimmune disease of the central nervous system and is a chronic and progressive disease characterized by inflammation, demyelination, and axonal degeneration. Due to axonal damage and demyelination, various neurological findings with motor and sensory losses are observed in patients with MS depending on their localization in the central nervous system. These findings vary depending on the location and size of the lesion, frequency, and severity of the disease. It is known that there are 2.8 million people living with MS in the world. Generally, the first symptoms appear between the ages of 20-40, but it is defined as early-onset or pediatric under the age of 18, adult-onset between the ages of 18-49, and late-onset after the age of 50. It is approximately twice as common in women, and is more common between the ages of 20-50, especially in white races. Although four clinical types are defined in MS: relapsing remitting MS, primary progressive MS, secondary progressive MS, relapsing progressive MS, clinically isolated MS has been added to the current classification, and the relapsing progressive MS classification has been abolished and those in this classification have been included in the primary progressive MS class. The relapsing remitting type is the most common, and there are periods of exacerbation (relapse) and remission in this type. Complications that occur during the exacerbation period show full or near-full recovery during the remission period. Various neurological findings such as spasticity, muscle weakness, gait disturbance, cognitive impairment, swallowing problems, bladder-bowel dysfunction can be observed in MS patients, and respiratory complications constitute one of the most common and important causes of death in MS. The risk of death is almost 12 times higher due to respiratory complications, which constitute approximately 47% of the causes of death in MS. Involvement of the pulmonary system, which is usually observed to have deterioration in diffusion capacity, respiratory muscle strength, and ventilation-perfusion ratio, leads to exercise intolerance, hospitalization, and mortality in MS. In MS, the primary factor is the formation of demyelinating plaques in the central nervous system, and the secondary factors include medications used, fatigue due to the disease, increased body temperature, a sedentary lifestyle, and loss of fitness, which all come together to cause pulmonary effects such as respiratory muscle weakness, lung volume deterioration, neurogenic pulmonary edema, sleep-disordered breathing, impaired respiratory control, decreased coughing efficiency, and respiratory failure. When the literature is examined, it seems that there is a need to try new methods in these disease groups to prevent respiratory complications and improve respiration due to pulmonary effects seen in MS. This study aims to investigate the effects of functional inspiratory muscle training, basic inspiratory muscle training, and physical activity applied in addition to respiratory exercises on respiratory muscle strength, respiratory function, cognitive function, walking, balance, functional exercise capacity, physical activity, quality of life, and core muscles in patients with Relapsing Remitting type Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Relapsing Remitting Type Multiple Sclerosis (RRMS),
* EDSS (Expanded Disability Status Scale in MS: EDSS) score ranging from 1-5,
* Able to communicate (speak, understand, read and understand Turkish),
* Individuals who have not had an attack in the last three months,
* Individuals who have not received respiratory-based rehabilitation in the last six months will be included in the study.

Exclusion Criteria:

* Those with neurological diseases other than MS,
* Those who have functional exercise restrictions,
* Those with chronic cardiac or pulmonary diseases such as chronic obstructive pulmonary disease (COPD), asthma, interstitial lung disease and heart failure that may affect respiratory muscle strength and respiratory functions,
* Individuals who have had pneumonia due to viral or bacterial infection in the last six months or COVID-19 positive individuals proven by PCR-RT,
* Those with orthopedic problems, persistent neck and back pain and/or radiculopathy that prevent them from participating in the study,
* Those with diagnosed psychiatric disorders,
* Those who use tobacco and tobacco products,
* Participants with cooperation problems that may prevent evaluations and treatment will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Inspiratory Respiratory Muscle Strength | 8 weeks
  Participants' respiratory muscle strength will be measured with a portable device (Micro Medical Micro RPM, UK) that can measure intraoral pressure electronically, which is a non-invasive method, and the results will be recorded as maximal inspiratory pressure (MIP). The participant's nose will be closed with a valve while they are maximally expiratory in a sitting position, and a maximal inspiration will be requested for 1 - 3 seconds to complete the MIP measurement and the measurements will be recorded. The highest of the three best results, with no more than 10% difference between them, among at least five measurements will be recorded as the final data.
Expiratory Respiratory Muscle Strength | 8 weeks
  Participants' respiratory muscle strength will be measured with a portable device (Micro Medical Micro RPM, UK) that can electronically measure intraoral pressure, which is a non-invasive method, and the results will be recorded as maximal expiratory pressure (MEP). MEP measurement will be completed by closing the nose of the participant who is maximally inspiratory in a sitting position with a valve and asking the participant to exhale maximally for 1-3 seconds, and the measurements will be recorded. The highest of the three best results, with no more than 10% difference between them, among at least five measurements will be recorded as the final data.
Respiratory Function (FEV₁) | 8 weeks
  Respiratory functions will be assessed with a portable spirometer with the patient in a sitting position according to the criteria set by the American Thoracic Society and the European Respiratory Society. Spirometry measures multiple parameters during a single test. Participants will be asked to take a single forced breath during normal breathing and then exhale a single forced breath, measuring the forced expiratory volume (FEV₁) in the first second of the lung function test.
Respiratory Function (FVC) | 8 weeks
  Participants will be asked to take a single forced breath during normal breathing and then exhale a single forced breath, measuring the forced vital capacity (FVC) of the lung function test.
Respiratory Function (FEV₁/FVC) | 8 weeks
  Participants will be asked to take a single forced breath during normal breathing and then exhale a single forced breath, measuring the forced expiratory volume in the first second/forced vital capacity ratio (FEV₁/FVC) of the lung function test.
Respiratory Function (PEF) | 8 weeks
  Participants will be asked to take a single forced breath during normal breathing and then exhale a single forced breath, measuring peak expiratory flow rate (PEF) of the lung function test.
Respiratory Function (FEF%25-75) | 8 weeks
  Participants will be asked to take a single forced breath during normal breathing and then exhale a single forced breath, measuring forced expiratory midflow rate (FEF%25-75) of the lung function test.
Respiratory Function (VC) | 8 weeks
  Respiratory function will be assessed with a portable spirometer with the patient in a sitting position according to the criteria determined by the American Thoracic Society and the European Respiratory Society. The test will be repeated three times. Participants will be asked to inhale deeply and exhale deeply for sixty seconds. As a result of three consecutive tests, the highest and percentages of the expected vital capacity (VC) values of respiratory function will be obtained.
Paced Auditory Serial Addition Test (PASAT) | 8 weeks
  PASAT test is a test used to evaluate attention, processing speed and working memory. Within the scope of the test, participants are required to add numbers given at a certain speed and add each new number to the previous number.
Symbol Digit Modalities Test (SDMT) | 8 weeks
  This test is a test that measures cognitive processing speed. Patients match the numbers corresponding to certain symbols by finding their equivalents as much as possible.
Stroop Test | 8 weeks
  The Stroop test will be used to measure executive functions and attention control. Participants are asked to name the ink colors of words written with color names. For example, when the word "green" is written in blue ink, participants should say "blue."
Walking | 8 weeks
  Participants' walking will be evaluated with a 10-meter walking test. Participants will be positioned at the starting line in a pre-measured 10-meter area and the time will be started when the participant steps on the starting line. If the participant uses a walking aid, they will be allowed to walk with it and the measurement will be made twice. The time will end when the participant crosses the finish line at the end of the 10 meters and the best value will be recorded in m/sec.
Balance | 8 weeks
  Balance will be evaluated with a timed up and go test. The participant, sitting on the chair, with feet flat on the floor and arms resting on the chair rest, will be asked to get up from the chair, walk the previously measured three-meter area at a safe and normal pace, turn, walk back, and sit back on the chair. The time will be measured in seconds for three repetitions and the best result will be recorded.
Functional Exercise Capacity | 8 weeks
  The functional exercise capacity of the participants will be measured with a 6-minute walk test. The 6-minute walk test is used to determine the maximum distance the participant can walk in six minutes. It is used to measure walking fatigue and walking endurance. Before starting the test, the participants will be informed that they will have to walk as fast as possible without running in a thirty-meter corridor for six minutes and that they can rest by taking a break if they wish, but their rest periods will not be added to the six minutes. The participants will be encouraged once per minute with standard expressions during walking. The distance the participant has walked at the end of the six minutes will be recorded in meters.
Physical Activity | 8 weeks
  Participants' physical activity status will be assessed with the International Physical Activity Questionnaire short form (SF-IPAQ). The survey consists of seven questions. The duration and frequency of each activity performed in the last week are questioned in the survey. The MET values defined for walking (3.3 METs), moderate-intensity physical activity (4.0 METs) and vigorous-intensity physical activity (8.0 METs) will be multiplied by duration (minutes) and frequency (days) to reach physical activity score values (MET-min/week).
Quality of Life | 8 weeks
  The participants' quality of life will be assessed with the Multiple Sclerosis International Quality of Life Questionnaire, a MS-specific assessment scale. The scale consists of nine subgroups; Daily Living Activities, Psychological Status, Findings, Relationships with Friends, Family Relations, Emotional and Sexual Life, Acceptance of the Disease, Coping with the Disease and Relationships with Medical Personnel. Each question in this scale, consisting of a total of 31 questions, is scored between 0-4 as "Never, Never" (0 points), "Rarely, A Little" (1 point), "Sometimes, A Little" (2 points), "Frequently, A Lot" (3 points), "Always, A Lot" (4 points). In the evaluation, the total score is calculated and the actual score is obtained by dividing by 1.24 for linear transformation, since the maximum score that can be obtained from the scale is 124. Low scores indicate high quality of life.
Core Muscles (Pelvic Bridge Test) | 8 weeks
  The pelvic bridge test and modified plank test will be used to assess the stabilization of the core muscles. For the pelvic bridge test, participants will be asked to lie on their backs with their knees flexed and their arms extended at their sides, and then they will be instructed to straighten their trunk by lifting their pelvic region. The time they can maintain this position will be recorded.
Core Muscles (Modified Plank Test) | 8 weeks
  The pelvic bridge test and modified plank test will be used to assess the stabilization of the core muscles. In the modified plank test, participants will be shown a series of movements and the time they maintain these positions will be recorded and measured.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail ÖZSOY, Assoc. Prof. Dr., Study Director — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Selen GUR OZMEN, Assoc. Prof. Dr., Study Director — Bahcesehir University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Istanbul, Türkiye
Locations (1):
- Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tong TK, Wu S, Nie J. Sport-specific endurance plank test for evaluation of global core muscle function. Phys Ther Sport. 2014 Feb;15(1):58-63. doi: 10.1016/j.ptsp.2013.03.003. Epub 2013 Jul 11. PMID 23850461
- [Background] Simeoni M, Auquier P, Fernandez O, Flachenecker P, Stecchi S, Constantinescu C, Idiman E, Boyko A, Beiske A, Vollmer T, Triantafyllou N, O'Connor P, Barak Y, Biermann L, Cristiano E, Atweh S, Patrick D, Robitail S, Ammoury N, Beresniak A, Pelletier J; MusiQol study group. Validation of the Multiple Sclerosis International Quality of Life questionnaire. Mult Scler. 2008 Mar;14(2):219-30. doi: 10.1177/1352458507080733. Epub 2007 Oct 17. PMID 17942521
- [Background] Shubert TE, Schrodt LA, Mercer VS, Busby-Whitehead J, Giuliani CA. Are scores on balance screening tests associated with mobility in older adults? J Geriatr Phys Ther. 2006;29(1):35-9. PMID 16630375
- [Background] Savcı, F. D. S., Öztürk, U. F. M., & Arıkan, F. D. H. (2006). Üniversite öğrencilerinin fiziksel aktivite düzeyleri. Türk Kardiyol Dern Arfl, 34(3), 166-172.
- [Background] Saglam M, Arikan H, Savci S, Inal-Ince D, Bosnak-Guclu M, Karabulut E, Tokgozoglu L. International physical activity questionnaire: reliability and validity of the Turkish version. Percept Mot Skills. 2010 Aug;111(1):278-84. doi: 10.2466/06.08.PMS.111.4.278-284. PMID 21058606
- [Background] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Background] Neder JA, Andreoni S, Lerario MC, Nery LE. Reference values for lung function tests. II. Maximal respiratory pressures and voluntary ventilation. Braz J Med Biol Res. 1999 Jun;32(6):719-27. doi: 10.1590/s0100-879x1999000600007. PMID 10412550
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Lin MR, Hwang HF, Hu MH, Wu HD, Wang YW, Huang FC. Psychometric comparisons of the timed up and go, one-leg stand, functional reach, and Tinetti balance measures in community-dwelling older people. J Am Geriatr Soc. 2004 Aug;52(8):1343-8. doi: 10.1111/j.1532-5415.2004.52366.x. PMID 15271124
- [Background] IPAQ Research Committee. (2005). Guidelines for data processing and analysis of the International Physical Activity Questionnaire (IPAQ)-short and long forms.
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Akuthota V, Ferreiro A, Moore T, Fredericson M. Core stability exercise principles. Curr Sports Med Rep. 2008 Feb;7(1):39-44. doi: 10.1097/01.CSMR.0000308663.13278.69. PMID 18296944
- [Background] McConnell, A. (2013). Respiratory muscle training: theory and practice. Elsevier Health Sciences.
- [Background] Dereli, M., Ozcan Kahraman, B., & Kahraman, T. (2022). A narrative review of respiratory impairment, assessment, and rehabilitation in multiple sclerosis. Dubai Medical Journal, 5(1), 78-88.
- [Background] Tzelepis GE, McCool FD. Respiratory dysfunction in multiple sclerosis. Respir Med. 2015 Jun;109(6):671-9. doi: 10.1016/j.rmed.2015.01.018. Epub 2015 Feb 12. PMID 25724874
- [Background] Hirst C, Swingler R, Compston DA, Ben-Shlomo Y, Robertson NP. Survival and cause of death in multiple sclerosis: a prospective population-based study. J Neurol Neurosurg Psychiatry. 2008 Sep;79(9):1016-21. doi: 10.1136/jnnp.2007.127332. Epub 2008 Feb 26. PMID 18303108
- [Background] Ascherio A, Munger KL. Environmental risk factors for multiple sclerosis. Part I: the role of infection. Ann Neurol. 2007 Apr;61(4):288-99. doi: 10.1002/ana.21117. PMID 17444504
- [Background] Klineova S, Lublin FD. Clinical Course of Multiple Sclerosis. Cold Spring Harb Perspect Med. 2018 Sep 4;8(9):a028928. doi: 10.1101/cshperspect.a028928. PMID 29358317
- [Background] Koch-Henriksen N, Sorensen PS. The changing demographic pattern of multiple sclerosis epidemiology. Lancet Neurol. 2010 May;9(5):520-32. doi: 10.1016/S1474-4422(10)70064-8. PMID 20398859
- [Background] Usta NC, Boz C, Terzi M. Early onset multiple sclerosis and the effect of disease onset age on neurological disability in multiple sclerosis. Clin Neurol Neurosurg. 2023 Jan;224:107528. doi: 10.1016/j.clineuro.2022.107528. Epub 2022 Nov 23. PMID 36446265
- [Background] Wilson S, Calocer F, Rollot F, Fauvernier M, Remontet L, Tron L, Vukusic S, Le Page E, Debouverie M, Ciron J, Ruet A, De Seze J, Zephir H, Moreau T, Lebrun-Frenay C, Laplaud DA, Clavelou P, Labauge P, Berger E, Pelletier J, Heinzlef O, Thouvenot E, Camdessanche JP, Leray E, Dejardin O, Defer G. Effects of socioeconomic status on excess mortality in patients with multiple sclerosis in France: A retrospective observational cohort study. Lancet Reg Health Eur. 2022 Nov 17;24:100542. doi: 10.1016/j.lanepe.2022.100542. eCollection 2023 Jan. PMID 36426377
- [Background] Brown TR, Kraft GH. Exercise and rehabilitation for individuals with multiple sclerosis. Phys Med Rehabil Clin N Am. 2005 May;16(2):513-55. doi: 10.1016/j.pmr.2005.01.005. PMID 15893685
- [Background] Bishop M, Rumrill PD. Multiple sclerosis: Etiology, symptoms, incidence and prevalence, and implications for community living and employment. Work. 2015;52(4):725-34. doi: 10.3233/WOR-152200. PMID 26639011
- [Background] Tremlett H, Paty D, Devonshire V. Disability progression in multiple sclerosis is slower than previously reported. Neurology. 2006 Jan 24;66(2):172-7. doi: 10.1212/01.wnl.0000194259.90286.fe. PMID 16434648
- [Background] Calabresi PA. Diagnosis and management of multiple sclerosis. Am Fam Physician. 2004 Nov 15;70(10):1935-44. PMID 15571060
- [Background] Filippi M, Bar-Or A, Piehl F, Preziosa P, Solari A, Vukusic S, Rocca MA. Author Correction: Multiple sclerosis. Nat Rev Dis Primers. 2018 Nov 22;4(1):49. doi: 10.1038/s41572-018-0050-3. PMID 30467372
- [Background] Centonze D, Leocani L, Feys P. Advances in physical rehabilitation of multiple sclerosis. Curr Opin Neurol. 2020 Jun;33(3):255-261. doi: 10.1097/WCO.0000000000000816. PMID 32304436